CLINICAL TRIAL: NCT05693623
Title: The Effect of Cold Application to the Sacral Area in the Transition Phase of Labor on Labor Comfort:
Brief Title: The Effect of Cold Application to the Sacral Area on Labor Comfort:
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Emine Yıldırım (Other)
Responsible Party: Sponsor-Investigator, Emine Yıldırım, Doktor Öğretim Üyesi, Osmaniye Korkut Ata University
Organization: Osmaniye Korkut Ata University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 12345
Record Dates: First submitted 2022-08-18; First posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Birth

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold Application to the Sacral Area (Experimental)
  Interventions: Other: cold application
- control group (No Intervention)

INTERVENTIONS:
Other: cold application — cold application
  Arms: Cold Application to the Sacral Area

SUMMARY:
Purpose: Cold application is considered as an effective alternative treatment for labor comfort because of its low side effects and easy availability. This study aims to determine the effect of cold application to the sacral area in the transition phase of labor on labor comfort.

Materials and methods: The study was done as a randomised controlled experimental study. While the women in the experimental group received cold application for 10 minutes every 20 minutes after 8 cm of cervical dilatation, the women in control group received routine care protocol of the unit.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were having a full-term pregnancy (pregnancies between 37th and 42nd weeks),
* having a single fetus, having a cephalic presentation,
* fetal weight of 2,5- 4 kg,
* pregnant women's having normal body mass index and receiving no antenatal trainings,
* having an 8 cm cervical dilation.

Exclusion Criteria:

* The women who had any kind of pregnancy complications (placenta previa, preeclampsia,
* premature rupture of membranes, oligohydramnios and polyhydramnios, presentation disorder,
* intrauterine growth retardation, intrauterine dead fetus,
* macrosomia babies, fetal distress, etc.),
* who had any systemic or neurologic diseases
* contraction anomalies (hypotonic or hypertonic contractions),
* who had induced labor,
* who received narcotic analgesics,
* who had occiput posterior,
* who were in the latent and active phases of labor,
* who had irregular contractions were excluded from the study

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-20 (Estimated); Primary Completion 2023-02-20 (Estimated); Study Completion 2023-03-20 (Estimated)

PRIMARY OUTCOMES:
Cold Application to the Sacral Area on Labor Comfort | through study completion, an average of 1 year
  Cold Application to the Sacral Area on Labor Comfort